CLINICAL TRIAL: NCT01251484
Title: Phase II Study of BIBF 1120 in Recurrent Glioblastoma Multiforme
Brief Title: BIBF 1120 in Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ulrik Lassen (Other)
Collaborators: Boehringer Ingelheim (Industry); University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Ulrik Lassen, Ulrik Lassen, MD, PH.D, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIBF1120 GBM
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: BIBF1120 — Tablet 200 mg twice daily until progression

SUMMARY:
VEGF inhibition by BEV may induce a change in tumor invasiveness and treatment failure is often associated with remote metastases. BEV may stop the growth of tumor cells by blocking blood flow to the tumor. Cediranib, a pan-VEGF inhibitor has shown promising results in recurrent GBM.

VEGF-blocking with small molecules may overcome the mechanism of resistance, and response to BIBF-1120 in such circumstances may open a new treatment option in GBM. In additional, recurrent glioblastomas have an extremely poor prognosis, so innovative therapies are needed.

ELIGIBILITY:
Inclusion criteria

* Written informed consent
* Histological verification of primary GBM and failure after radiotherapy and TMZ

  - Previously received radiotherapy and TMZ
* More than 4 weeks since any of the following prior treatments

  * Chemotherapy (6 weeks for nitrosureas or mitomycin C)
  * Radiotherapy to nontarget lesions or lesions that are not to be biopsied
  * Investigational agents
* More than 6 months since prior major surgery or open biopsy and recovered (only 6 weeks required if operation is for recurrent BGM)
* ● ECOG performance status 0-1
* Age > 18 years
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Fertile females must use anticonception (p- pills, IUD, depot injection of gestagen, subdermal
* implantation, hormonal vaginal ring or transdermal depot plaster, throughout the study and 3
* months after discontinuation of study drugs. Fertile men must use dobbelt barrier method
* (preservative with sperm inhibiting creme) or female partner uses the above mentioned
* contraception.
* Fertile males must use preservatives.

Exclusions criteria

* Prior treatment with BIBF 1120 or any other VEGFR inhibitor, except bevacizumab in Group 2
* Chemo-, hormono-, radio-(except for brain and extremities) or immunotherapy or therapy with monoclonal antibodies or small tyrosine kinase inhibitors within the past 4 weeks prior to treatment with the trial drug.
* Persistence of clinically relevant therapy related toxicity from previous chemo and/or radiotherapy
* Treatment with other investigational drugs or treatment in another clinical trial within the past 4 weeks before start of therapy or concomitantly with the trial
* Therapeutic anticoagulation( except low-dose heparin and/or heparin flush as needed for maintenance of an in-dwelling intravenous devise) or anti-platelet therapy (except for low-dose therapy with acetylsalicylic acid<325mg per day
* Major injuries within the past 10 days prior to start of study treatment with incomplete wound healing and/or planned surgery during the on-treatment study period
* History of clinically significant haemorrhagic or thromboembolic event in the past 6 months
* Known inherited predisposition to bleeding or thrombosis
* Significant cardiovascular diseases ( i.e. uncontrolled hypertension, unstable angina, history of infarction within the past 12 months prior to start of study treatment, congestive heart failure > NYHA II, serious cardiac arrhythmia, pericardial effusion)
* Proteinuria CTCAE grade 2 or greater
* Hepatic function: total bilirubin outside of normal limits; ALT or AST > 1.5 ULN
* Coagulation parameters: International normalised ratio ( INR) > 2, prothrombin time

  - (PT) and partial thromboplastin time (PTT) > 50% of deviation of institutional ULN
* Absolute neutrophil count ( ANC) < 1500/ml, platelets < 100000/ml, Haemoglobin < 9.0 g/dl
* Other malignancies within the past 5 years other then basal cell skin cancer or carcinoma in situ of the cervix
* Active serious infections in particular if requiring systemic antibiotic or antimicrobial therapy
* Active or chronic hepatitis C and/or B infection
* Gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug
* Serious illness or concomitant non-oncological disease such as neurologic, psychiatric, infectious disease or active ulcers (gastro-intestinal tract, skin) or laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the study.
* Pregnancy or breast feeding
* Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule
* active alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Response rate | Response evaluation every 8 weeks
  MacDonald criteria

SECONDARY OUTCOMES:
Adverse events | Assessed every 2 weeks
  CTCAE version 4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark